CLINICAL TRIAL: NCT06148844
Title: The Effect of Interactive Robot on Pre-operative Anxiety and Fear of Children
Brief Title: Interactive Robot on Pre-operative Anxiety and Fear of Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karamanoğlu Mehmetbey University (Other)
Responsible Party: Principal Investigator, Tuba Arpacı, Asisstant Professor, Karamanoğlu Mehmetbey University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: KMU-SBF-TA-01
Record Dates: First submitted 2023-11-20; First posted 2023-11-28 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Surgery
Keywords: minor surgical procedures; nursing; interactive robot; chlidren

STUDY DESIGN:
Intervention Model Description: Two group with conventional therapy control group
Who Masked: Participant, Outcomes Assessor
Masking Description: Control group will receive conventional pre-operative preparation and intervention group will receive pre-operative preparation designed with interactive robot by researchers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): The routine preparation procedure in this group in the hospital will be applied by the nurses responsible for preoperative preparation. After pre-operative preparation, the child, parent and nurse will be asked to fill out the anxiety and fear scales to evaluate the child's anxiety and fear levels.
- Interactive robot group (Experimental): In addition to the routine preparation procedure interactive robot will be used to preparation as a therapeutic approach. The interactive robot will accompany to the child the preparation for the surgery. Then, the features of the interactive robot will be explained to the children and parents and it will be introduced to the children. The interactive robot will meet the child with its speech feature and the robot will accompany to child to the operating room entrance. The child will be informed that he/she can request the interactive robot to follow him/her if he/she wishes. The child will be transferred to the operating room accompanied by the nurse, researcher and robot. After pre-operative preparation, the child, parent and nurse will be asked to fill out the anxiety and fear scales to evaluate the child's anxiety and fear levels.
  Interventions: Other: interactive robot group

INTERVENTIONS:
Other: interactive robot group — Intervention group will receive one day pre-operative preparation intervention applied by researcher. Preparation will be 30-40 minutes long
  Arms: Interactive robot group

SUMMARY:
The aim of this study is to determine the effect of preoperative preparation applied with an interactive robot on children's preoperative anxiety and fear levels.

Hypothesis;

H1: Pre-operative preparation with an interactive robot has an effect on the anxiety level of children H2: Pre-operative preparation with an interactive robot has an effect on the fear level of children H3: The anxiety levels of children in intervention and control groups are different after the pre-operative preparation H4: The fear levels of children in intervention and control groups are different after the pre-operative preparation

DETAILED DESCRIPTION:
The use of interactive robots can be preferred as a remarkable method of communication with hospitalized children. In this way, it will be easier for the children to understand the procedure and they will be able to communicate easily with healthcare professionals. Children may develop a sense of control and the level of anxiety and fear they experience may decrease when they interact with robots. It is reported in the literature that children show more interest in robots than they do in adults. In addition, children see social robots as living creatures, not as devices, and children who spend time with them for a long time adopt them as friends. In a study, a social humanoid robot was used to prepare children aged 7-12 (n = 11) regarding the cancer diagnosis process and interventional procedures. According to the results of the study, the children's stress, depression, and anger during the treatment decreased significantly. Interactive robots positively affect postoperative mobilization in children undergoing day surgery and reduce the anxiety level of children before mobilization. As a result, it may be easier for children to cope with stress with the use of interactive and humanoid robots. Also, interactive robots can facilitate cooperation between the child and the nurse by playing an intermediary role in communication with children. Determining the effects of interactive robots on children by using them before the surgical procedure is important to ensure the active participation of children in the surgical process in pediatric surgery clinics. It is thought that this research is important in terms of interventions which appropriate to the supportive care role of nurses and will contribute to the literature.

ELIGIBILITY:
Inclusion Criteria:

* Those between the ages of 5-10,
* having planned day surgery,
* scheduled for general anesthesia
* have not had surgery before,
* Those who can speak Turkish

Exclusion Criteria:

* Children have mental-cognitive problems,
* Children have hearing, vision and/or speech disabilities

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 74 (Actual)
Dates: Start 2023-09-18 (Actual); Primary Completion 2023-11-18 (Actual); Study Completion 2023-11-18 (Actual)

PRIMARY OUTCOMES:
Anxiety | one day
  Children's State Anxiety Scale: Validated scale used for evaluation of 4-10 aged children's anxiety level. Scale score ranges between 0-10.
Fear | one day
  Children's Fear Scale: Validated scale used for evaluation of 5-10 aged children's fear level. Scale score ranges between 0-4.

CONTACTS AND LOCATIONS:
Overall Officials: Tuba ARPACI, PhD, Principal Investigator — Karamanoğlu Mehmetbey University
Locations (1):
- Karaman Education and Research Hospital, Karaman, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No